CLINICAL TRIAL: NCT05760482
Title: Evaluation of the Relationship Between Bruxism and Tryptophan Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SelcukU002
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Bruxism; Anxiety State; Tryptophan Metabolism Alterations
MeSH Terms: conditions — Bruxism; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bruxism Group (Experimental)
  Interventions: Diagnostic Test: Metobolites serum level measurement; Behavioral: Anxiety and stress level measurement
- Control Group (Experimental)
  Interventions: Diagnostic Test: Metobolites serum level measurement; Behavioral: Anxiety and stress level measurement

INTERVENTIONS:
Diagnostic Test: Metobolites serum level measurement — Blood samples will be taken from all volunteer participants in 1 yellow cap tube of 10 cc. After the blood has cooled and the clot development process (approximately 15 minutes), the serum will be separated by centrifugation at 2000 g for 5 minutes. Separated sera will be aliquoted and stored at -40°C until analysis. The tryptophan and tryptophane metabolite levels of the participants will be measured by Liquid Chromatography-Tandem Mass Spectrometer API 3200 device. The kynurenine, kynurenic acid, 3-HK, 3-HAA, 3-HOA, and QA values obtained as a result of this test will be recorded.
Behavioral: Anxiety and stress level measurement — Anxiety and stress levels will be evaluated by applying State-Trait Anxiety Inventory and Perceived Stress Scale Tests by all volunteer participants. Scores from these tests will be recorded.

SUMMARY:
Psychological causes are often cited as the most important of the underlying factors for bruxism. However, there are very few studies that can objectively demonstrate this. There are studies that are generally based on subjective data, that is, on questionnaires that indicate anxiety or stress. Recent studies have shown that tryptophan and its metabolites are associated with psychological health. In this study, researchers will measure the serum values of metabolites in the tryptophan pathway. Also, researchers will observe whether these metabolite levels differ significantly in patients with and without bruxism.

DETAILED DESCRIPTION:
Bruxism is a common health problem that occurs throughout life and has a prevalence of 9% to 31% among adults. This common muscle disorder, characterized by teeth grinding or clamping, which can occur during sleep or day, is considered multifactorial with potential effects on the central nervous system. A possible relationship between mental health and bruxism has been investigated due to the indication of psychological factors such as anxiety and stress at the onset of bruxism. It has been reported that when the presence of mental disorders causes changes in the regulation of the central nervous system, they can act as a trigger point for bruxism.

Depression and anxiety disorders are the most common mental disorders studied and are expected to be the most common chronic condition by 2050. The emerging field of nutritional psychiatry offers some opportunities for clinical intervention for individuals suffering from depression and anxiety. L-tryptophan, a precursor of serotonin, is expected to contribute to the correction of depressive and anxious moods.

The primary catabolic pathway of tryptophan is the pathway of kynurenine, which is responsible for about 95-99% of tryptophan metabolism in the body. Tryptophan turns into kynurenine in the kynurenine pathway and is divided into two pathways. The first forms kynurenic acid, while the other forms 3-hydroxykynurenine (3-HK), 3-hydroxyanthranylic acid (3-HAA), and quinolinic acid (QA), respectively. The first pathway is considered neuroprotective, while the second pathway is known as neurotoxic.

In studies trying to explain the link between tryptophan and its metabolites and depression, they have emphasized that depression is caused by an imbalance in the kynurenine pathway and that the amount of quinolinic acid, which is neurotoxic, increases, while peripheral kynurenine, which is neuroprotective, decreases. It has been shown that the neurotoxic metabolites formed in the kynurenine itself and its pathway may be associated with depression and anxiety. There are researchers who think that changes in these parameters and their proportions to each other indicate different psychological states.

Changes in serum levels of these metabolites in cases of stress and anxiety have been supported by the studies mentioned above. Although most authorities assume that bruxism is based on psychological factors, the studies supporting them are usually anxiety and stress-focused survey studies based on subjective data. This assumption; researchers could not find a study comparing it with objective data. This study aims to present a possible relationship between bruxism and tryptophan metabolites in volunteer individuals with and without bruxism. The researchers' initial hypothesis is that "Changes in tryptophan and catabolites play a role in the etiology of bruxism."

ELIGIBILITY:
Inclusion Criteria:

* age range 18-50
* applying to our clinic with the complaint of bruxism
* no psychological drug
* no active orthodontic treatment
* no musculoskeletal disease
* no removable prosthesis
* no obstructive sleep apnea syndrome
* "Class I" according to RDC/TMD classification
* "probable" according to bruxism classifiacation
* accept to fill out the questionnaire
* accept to give a blood sample
* being volunteer
* accept to sign the informed consent

Exclusion Criteria:

* indicate to quit the study at anytime
* not fully fill out the questionnaire
* encountering any complication during taking a blood sample
* can not take an adequate blood sample
* presenting any below diseases;

  1. acute myocardial infarction
  2. pulmonary emboli
  3. deep venous thrombosis
  4. heart failure
  5. sepsis
  6. cerebral edema
  7. hypertensive encephalopathy
  8. hypoglycemia
  9. hepatic encephalopathy
  10. fluid-electrolyte disturbances
  11. acute-chronic renal failure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
serum tryptophane level measurement | blood sample will be taken 5 minutes after the patient sits the dental unit
  serum tryptophane level measurement
serum kynurenin level measurement | blood sample will be taken 5 minutes after the patient sits the dental unit
  serum kynurenin level measurement
serum kynurenic acid level measurement | blood sample will be taken 5 minutes after the patient sits the dental unit
  serum kynurenic acid level measurement
serum quinolinic acid level measurement | blood sample will be taken 5 minutes after the patient sits the dental unit
  serum quinolinic acid level measurement
serum 3-hydroxykynurenin level measurement | blood sample will be taken 5 minutes after the patient sits the dental unit
  serum 3-hydroxykynurenin(3-HK) level measurement
serum 3-hydroxyanthranilic level measurement | blood sample will be taken 5 minutes after the patient sits the dental unit
  serum 3-hydroxyanthranilic(3-HAA) level measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Gürses, Assistant Professor, Study Chair — Selcuk University, Faculty of Dentistry; Ali Ünlü, Professor, Principal Investigator — Selcuk University, Faculty of Medicine
Locations (1):
- Selcuk University, Faculty of Dentistry, Konya, Selçuklu, Turkey (Türkiye)